CLINICAL TRIAL: NCT03434821
Title: Impact of Hyperoxemia on Incidence of Ventilator-associated Pneumonia
Brief Title: Hyperoxemia and Ventilator-associated Pneumonia
Acronym: SOH-VAP
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2016_73; 2017-A01934-49 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2018-02-06; First posted 2018-02-15 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Mechanical Ventilation
Keywords: Hyperoxemia; ventilator-associated; pneumonia; critical illness
MeSH Terms: conditions — Pneumonia; Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this prospective cohort single-center observational study is to determine the impact of hyperoxemia on ventilator-associated pneumonia (VAP) occurrence.

* SpO2 will be continuously recorded in order to determine the percentage of time spent with hyperoxemia.
* Patients with VAP will be prospectively identified.
* Patient characteristics and risk factors for VAP will be prospectively collected.
* Oxidant stress will be prospectively investigated in study patients: glutathion peroxidase (GPX), plasmatic superoxyde dismutase (SOD), total plasmatic antioxidant status (SAT) and urinary 8-isoprostanes will be performed at ICU admission, once a week, and at VAP occurrence.

Patients with VAP will be compared with those with no VAP

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to the ICU
* Expected duration of mechanical ventilation > 48h
* Signed informed consent
* Social insurance

Exclusion Criteria:

* Pregnancy or breast feeding
* No informed consent
* Hyperbaric oxygen treatment
* Prisoners and patients under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients hospitalized in intensive care unit requiring invasive mechanical ventilation (IV) for more than 48 hours.
Sampling Method: Non-Probability Sample
Enrollment: 534 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
VAP occurrence | 28 days after ICU admission
  hyperoxemia at ICU admission (PaO2 >120 mmHg)

SECONDARY OUTCOMES:
percentage of time spent with hyperoxemia during ICU stay | 28 days after ICU admission
  hyperoxemia is defined as peripheral O2 saturation (SaO2)>98%, SaO2 will be measured every 30 seconds, and the percentage of time spent with hyperoxemia will be calculated per day.
relationship between hyperoxemia at ICU admission and the presence of acute lung injury (ALI) | 28 days after ICU admission
  the presence of hyperoxemia at ICU admission will be determined using blood gazes (arterial PaO2>120 mmHg). The percentage of patients with hyperoxemia will be compared between patients with Ali, and those with no ALI
percentage of time spent with hyperoxemia during ICU stay, and the presence of acute lung injury | 28 days after ICU admission
  the percentage of time spent with hyperoxemia during ICU stay will be calculated as mentioned above (outcome 2). This percentage will be compared between patient with ALI and those with no ALI

CONTACTS AND LOCATIONS:
Overall Officials: Saad Nseir, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHU de Lille, Lille, France